CLINICAL TRIAL: NCT04812444
Title: Safety and Efficacy of Peripheral Venous Stent System in the Treatment of Patients With Iliac Vein Stenosis or Occlusion: a Prospective, Multicentre, Randomized Controlled Clinical Trial.
Brief Title: Peripheral Venous Stent System in the Treatment of Iliac Vein Stenosis or Occlusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang Zylox Medical Device Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZYLOX-02
Record Dates: First submitted 2020-11-03; First posted 2021-03-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Iliac Vein Stenosis; Iliac Vein Occlusion
Keywords: Peripheral venous stent system; Iliac vein patency rate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zylox Peripheral Venous Stent Implantation (Experimental): Percutaneous stent placement in the iliofemoral veins
  Interventions: Device: Zylox Peripheral Venous Stent
- Zilver Vena Venous Stent Implantation (Active Comparator): Percutaneous stent placement in the iliofemoral veins
  Interventions: Device: Zilver Vena Venous Stent

INTERVENTIONS:
Device: Zylox Peripheral Venous Stent — Self-expanding stent implantation during the index procedure.
  Arms: Zylox Peripheral Venous Stent Implantation
Device: Zilver Vena Venous Stent — Self-expanding stent implantation during the index procedure.
  Arms: Zilver Vena Venous Stent Implantation

SUMMARY:
Clinical study on safety and efficacy of Zylox peripheral venous stent system in the treatment of iliac vein stenosis or occlusion.

DETAILED DESCRIPTION:
The purpose of this study was to evaluate the safety and efficacy of Zylox peripheral venous stent system in the treatment of iliac vein stenosis or occlusive lesions compare with conventional venous stent.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 18 to 75 years old, male or female
* Subject's target lesions were stenosis and/or occlusion
* CEAP≥C3
* Subjects were able to understand the purpose of the study, demonstrate full compliance with the program and sign informed consent

Exclusion Criteria:

* Pregnant woman or who's pregnancy test is positive
* Lactation period woman or woman/man with fertility plan

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2020-10-09 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
Target vascular patency rate at 12 months after operation | 12 months
  Target vascular patency rate

SECONDARY OUTCOMES:
The incidence of major adverse events | 12 months
  Related to death of clinical trials
Adverse Event | Preoperative、Intraoperative、up to 1 month、3 month、6 month、12 month、2 years、3 years、5 years
  Adverse medical events,whether or not related to the medical device

CONTACTS AND LOCATIONS:
Overall Officials: Yu Zhao, Principal Investigator — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China